CLINICAL TRIAL: NCT05078398
Title: Postoperative Opt-In Narcotics Treatment in Breast
Acronym: POINT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, James Wu, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#21-001169
Record Dates: First submitted 2021-09-21; First posted 2021-10-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Surgery; Opioid Use
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POINT-B (Experimental): Patients will receive perioperative counseling on opioid consumption following breast surgery, both preoperatively and postoperatively. Upon discharge, patients will be asked whether they would like to be discharged with narcotic pain medication or not.
  Interventions: Behavioral: POINT Protocol
- Usual Care (Active Comparator): Patients will receive equivalent of 5 tabs of Norco 5/325 mg upon discharge routinely
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: POINT Protocol — Patients will receive counseling on risks and benefits of opioids for pain control, asked to choose whether they need opioid prescription when ready for discharge.
  Arms: POINT-B
Behavioral: Usual care — Will prescribe standardized amount of opioid for postoperative pain without patient input
  Arms: Usual Care

SUMMARY:
In a recent study, researchers let patients choose what medications to go home with after endocrine surgery. This has not been done in outpatient breast surgery, though several institutions have moved towards avoiding opioids altogether after breast surgery. These institutions only prescribed rescue opioids upon request.

The aim of this study is to compare a similar "opt-in" protocol for narcotics to usual care (where patients are routinely discharged with opioids) for outpatient breast surgery.

This study will be designed as a randomized, controlled trial. When adult patients consent for outpatient breast surgery, the patients will be asked to participate in the study. Patients who are currently using narcotics would be excluded. The investigators would then randomize participants to the "opt-in" protocol versus being provided with a standard opioid prescription after surgery. Patients in the opt-in protocol will be recommended a pain treatment regimen with over-the-counter medications, acetaminophen or ibuprofen. These patients will be reassured that if their pain is uncontrolled after discharge, a narcotic prescription will be called in to their pharmacy if requested.

The investigators will assess patient pain scores and medication use in the recovery area using the electronic medical record. The investigators will collect data on patient pain scores and medication use after discharge on a daily basis via phone call or electronically transmitted survey. The investigators will also evaluate patients at the time of their follow-up visits. Any patient phone calls will be routed to study personnel who will fill narcotic prescription requests if requested. Finally, among patients who do receive an opioid prescription, the investigators will track their opioid consumption.

DETAILED DESCRIPTION:
Due to the current opioid epidemic, there has been increased focus on the prescribing patterns of physicians and greater incentive to reduce the amount of narcotic pain medication prescribed.

A recent publication in Journal of American Medical Association Surgery conducted by researchers from the same institution found that giving patients the option of choosing to receive a narcotic prescription or not following endocrine surgery significantly reduced opioid prescriptions and waste without increased pain or worse quality of life. No patients called in to request narcotic pain medication after discharge.

Significance:

Given the current health care and political climate, there has been increasing focus on reducing the amount of narcotics prescribed by health care providers. Based on the results of the above cited study, the investigators believe implementing an opt-in program at University of California at Los Angeles will also significantly decrease the amount of opioids prescribed for postoperative pain following outpatient breast surgery as well.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing outpatient breast surgery (less than 24 hour stay)
* Understands written English

Exclusion Criteria:

* Current ongoing opioid use
* Increased complexity of surgery requiring longer hospital stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Daily peak pain scores on an 11-point numeric rating scale [0-10, with 0 indicating no pain and 10 indicating worst pain possible] | Postoperative day 0-7
  Daily peak pain
Number of opioid pills dispensed | Postoperative day 0-7
  Total number of pills, (also to be expressed in morphine equivalents) dispensed on day of surgery as well through the immediate post operative period if refills or a rescue prescription were requested

SECONDARY OUTCOMES:
Physical and Mental Health Summary Score from Patient-Reported Outcomes Measurement Information System (PROMIS) Survey (T-score, mean is 50 and 10 is standard deviation) | Baseline and postoperative day 7
  PROMIS Quality of life
Amount of opioid pills consumed | Postoperative day 0-7
  Total number of opioid pills consumed by patients during the immediate postoperative period (also to be expressed in morphine equivalents)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UCLA Santa Monica Medical Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: Undecided